CLINICAL TRIAL: NCT02831244
Title: Agili-CTM Implant Performance Evaluation in the Treatment of Osteoarthritis of the Great Toe
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Smith & Nephew, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLN0023
Record Dates: First submitted 2016-06-29; First posted 2016-07-13 (Estimated); Last update posted 2025-03-06 (Actual); Status verified 2020-02

CONDITIONS: Osteoarthritis of Multiple Joints of Ankle or Foot

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Agili-CTM (Other): Intervention
  Interventions: Device: Agili-CTM

INTERVENTIONS:
Device: Agili-CTM — Consenting individuals will be selected from the population of patients with osteoarthritis of the great toe examined by a participating investigator. Following signing an informed consent, candidates will be evaluated by an adjudication committee for possible inclusion in the trial based on medical history and Standing Foot X-ray. Candidates that are approved or conditionally approved by the adjudication committee will undergo Agili-CTM implantation procedure

SUMMARY:
The purpose of this study is to evaluate the performance of the Agili-CTM implant in the treatment of osteoarthritis of the Great Toe.

DETAILED DESCRIPTION:
Agili-C™ implant is a CE marked. The Agili-CTM implant is a porous resorbable tissue regeneration scaffold for the treatment of articular cartilage and/or osteochondral defects.

The Agili-C™ implant will be implanted using the Agili-Kit™ surgical toolset which is designed for the precise preparation of sites in cartilage and osteochondral defects, for implanting the Agili-C™ implant.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Osteoarthritis of the First Metatarsophalangeal Joint
* Presence of good bone stock
* Physically and mentally willing and able to comply with post-operative
* rehabilitation and routinely scheduled clinical and radiographic visits

Exclusion Criteria:

* < 18 years of age
* Any past or present evidence of infection of the treated joint
* Any known malignant tumor of the foot
* Known inflammatory arthropathy or crystal-deposition arthropathy
* Chemotherapy treatment in the past 12 months
* History of allergic reaction or intolerance to calcium carbonate or hyaluronate
* Patient who is pregnant or intends to become pregnant during the study
* History of any significant systemic disease, such as but not limited to, HIV infection, hepatitis infection or HTLV infection; known coagulopathies, that might compromise the subject's welfare
* Known substance abuse or alcohol abuse
* Participation in other clinical trials in parallel to this study
* Known insulin dependent diabetes mellitus
* Unable to undergo imaging studies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-08-10 (Actual); Primary Completion 2019-06-23 (Actual); Study Completion 2019-06-23 (Actual)

PRIMARY OUTCOMES:
Foot and Ankle Ability Measure (FAAM) score | 24 month
  FAAM score will be evaluated at 24 months compared to baseline
Visual Analog Scale (VAS) Pain | 24 month
  VAS will be evaluated at 24 months compared to baseline

SECONDARY OUTCOMES:
Great toe range of motion | 2 weeks, 6 weeks, 3, 6, 12 18 and 24 months
  Great toe range of motion will be evaluated at 2 weeks, 6 weeks, 3, 6, 12, 18 and 24 months compared to baseline
Pain according to Visual Analog Scale (VAS) | 2 weeks, 6 weeks, 3, 6, 12 and 18 months
  VAS score will be evaluated at 2 weeks, 6 weeks, 3, 6, 12 and 18 months
Activities of Daily Living Subscale according to Foot and Ankle Ability Measure (FAAM) | 2 weeks, 6 weeks, 3, 6, 12 and 18 months
  FAAM score will be evaluated at 2 weeks, 6 weeks, 3, 6, 12 and 18 months
AOFAS Hallux Metatarsophalangeal-Interphalangeal Scale (HMIS) score (American Orthopaedic Foot and Ankle Society-AOFAS) | 2 weeks, 6 weeks, 3, 6, 12, 18 and 24 months
  AOFAS will be evaluated at 2 weeks, 6 weeks, 3, 6, 12, 18 and 24 months compared to baseline
Measurament of Joint Space maintenance in mm | 12 and 24 months
  Joint Space maintenance will be evaluated at 12, and 24 months compared to baseline
Quality of life questionnaire (SF-36) | 6, 12, 18 and 24 months
  SF-36 will be evaluated at 6,12, 18 and 24 months compared to baseline

CONTACTS AND LOCATIONS:
Locations (4):
- Hasharon Medical Center, Petah Tikva, Israel
- Rizzoli Orthopedic Institute, Bologna, Italy
- Clinical Center of Vojvodina, Novi Sad, Serbia
- University Medical Centre, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Drobnic M, Vannini F, Kon E, Dulic O, Kecojevic V, Andor B, Altschuler N, Robinson D. Treatment of hallux rigidus by a novel bi-phasic aragonite-based implant: results of a two year multi-centre clinical trial. Int Orthop. 2021 Apr;45(4):1033-1041. doi: 10.1007/s00264-020-04872-8. Epub 2020 Nov 12. PMID 33184685